CLINICAL TRIAL: NCT05937295
Title: FusionVAC22_01: DNAJB1-PRKACA Fusion Transcript-based Peptide Vaccine Combined with Immune Checkpoint Inhibition for Fibrolamellar Hepatocellular Carcinoma and Other Tumor Entities Carrying the Oncogenic Driver Fusion
Brief Title: FusionVAC22_01: Fusion Transcript-based Peptide Vaccine Combined with Immune Checkpoint Inhibition
Acronym: FusionVAC22
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FusionVAC22_01; 2022-502869-17-01 (Other: Eu-CT Number)
Record Dates: First submitted 2023-05-09; First posted 2023-07-10 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Fibrolamellar Hepatocellular Carcinoma
Keywords: FL_HCC; DNAJB1-PRKACA
MeSH Terms: conditions — Fibrolamellar hepatocellular carcinoma

STUDY DESIGN:
Intervention Model Description: Phase I, open-label, multicenter, interventional clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FusionVAC-XS15 and Atecolizumab treatment (Experimental)
  Interventions: Drug: Fusion-VAC-XS15

INTERVENTIONS:
Drug: Fusion-VAC-XS15 — FusionVAC-22 peptide will be administered subcutaneously (s.c.) adjuvanted with the Toll-like receptor 1/2 ligand XS15 (50 μg) emulsified in Montanide ISA 51 VG (1:1).
  Vaccination will take place every 4 weeks at the beginning of Cycle 1 and 2. A total of two vaccinations are planned.
  After 11 months a booster vaccination can be applied depending on T-cell responses.
  Immune checkpoint inhibition (ICI):
  Atezolizumab (TecentriqTM, Roche Pharma AG) is a humanized immunoglobulin (Ig) G1 monoclonal antibody that targets PD-L1 and will be applied intravenously (i.v.).
  The anti-PD-L1 antibody Atezolizumab (TecentriqTM) 1680 mg will be applied every 4 weeks as a 30-minute infusion (60-minute first dose) starting on day 15 after the first vaccination. Anti-PD-L1 treatment will be continued after the end of vaccination phase throughout the complete study period until End of Treatment (EOT) or until disease progression or other reasons for study termination.

SUMMARY:
The aim of this clinical trial is to evaluate the immunogenicity along with safety and toxicity as well as first efficacy of a DNAJB1-PRKACA fusion transcript-based peptide vaccine (Fusion-VAC-XS15) in combination with anti-programmed cell death-ligand 1 immune checkpoint inhibition (ICI) by Atezolizumab (TecentriqTM) in patients with Fibrolamellar hepatocellular carcinoma (FL-HCC) or other cancer entities carrying the DNAJB1-PRKACA fusion transcript.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign a written informed consent document.
* Histologically confirmed FL-HCC or other malignant disease that is locally advanced or metastatic.
* Non-FL-HCC patients can be included

  * in case of disease progression after therapy and fulfilling at least one of the following criteria: i. no further standard therapy is available. ii. patient is considered unsuitable for further available standard therapy. iii. patient is unwilling to receive treatment with available standard therapy.
  * if no standard therapy exists.
* Presence of DNAJB1-PRKACA fusion transcript, assessed by RNA-based next-generation sequencing (NGS) or realtime-polymerase chain reaction amplification (RT-PCR).
* Age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Patients must have measurable disease per iRECIST (Response Evaluation Criteria in Solid Tumours).
* Negative SARS-CoV-2 rapid antigen test (as long as World Health Organization declares pandemic spread of SARS-CoV-2).
* Adequate organ function laboratory values

  1. Absolute Lymphocyte Count > 500/μl
  2. Platelets > 50.000/μl
  3. Creatinine clearance glomerular filtration rate > 30 ml/min
  4. Liver function Child-Pugh index class A or B7
  5. Alanine aminotransferase (ALT) and aminotransferase (AST) ≤ 5 times upper limit range
  6. Bilirubin ≤ 3 mg/dl
* Negative serological Hepatitis B test or negative PCR in case of positive serological test without evidence of an active infection, negative testing of Hepatitis C RNA, negative HIV test within 6 weeks prior to study inclusion.
* Female patients of child bearing potential (FCBP) and male patients with partners of child bearing potential, who are sexually active, must agree to the use of two effective forms (at least one highly effective method) of contraception. This should be started from the signing of the informed consent and be continued until 5 months (both female and male patients) after last dose of an Atezolizumab (TecentriqTM) or vaccination.
* For FCBP two negative pregnancy tests (sensitivity of at least 25 mIU/mL) prior to first application of a study drug (vaccination at visit V1), one at screening and the other one at visit V1 prior (<24h) to first vaccination.
* Postmenopausal or evidence of non-child-bearing status.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Unwilling or unable to follow the study schedule for any reason.
* Chemotherapy or other systemic therapy or radiotherapy, up to 14 days prior to the first dose of study drug.
* Concurrent or previous treatment within 30 days in another interventional clinical trial with an investigational anticancer therapy or any other investigational therapy, which would interfere with the study's primary and secondary endpoints.
* Major surgery within 28 days of dosing of study drug.
* Have not recovered from adverse events to grade ≤ 2 or baseline due to previous agents administered excluding alopecia and neurotoxicity (≤ 2 grade).
* History of autoimmune phenomena due to treatment with immunotherapy agents (including, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4 antibodies, etc.) (≥ grade 3).
* Treatment with immunotherapy agents (including, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4 antibodies, etc.) within 28 days prior of dosing of study drug.
* Have received any live vaccine within 28 days prior to study treatment.
* Known sensitivity to or history of allergic reactions to any of the investigational drugs or known hypersensitivity to Chinese hamster ovary cell products.
* History of severe allergic anaphylactic reactions to chimeric, human or humanized antibodies, or fusion proteins.
* Has active autoimmune disease that requires or has required systemic immunosuppressive treatment in the past 2 years.
* Presence of any tissue or organ allograft, regardless of need for immunosuppression, including corneal allograft. Patients with a history of allogeneic hematopoietic stem cell transplant will be excluded.
* Has a diagnosis of immunodeficiency.
* Systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 7 days prior to study drug administration.
* Symptomatic interstitial lung disease.
* Active or untreated brain metastases or leptomeningeal metastases.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, different metastatic cancer than the one leading to study enrollment, or psychiatric illness/social

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
To assess immunogenicity in terms of induction of peptide specific T-cell responses | through study completion, an average of 1 year
  The percentage of patients with an induction of T-cell response until 28 days after second vaccination will be the primary endpoint for efficacy. Peptide stimulated Peripheral Blood Mononuclear Cells (PBMCs) are analyzed by enzyme-linked immunospot (ELISPOT).
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of the peptide vaccine in combination with anti-PD-L1 immune checkpoint inhibition | through study completion, an average of 1 year
  The safety and toxicity of the personalized multi-peptide vaccine in combination with the toll-like receptor1/2 ligand XS15 with anti-PD-L1 immune checkpoint inhibition (ICI) will be determined based on the Common Terminology Criteria for Adverse Events (CTCAE version 5.0) and assessed in a descriptive manner.

CONTACTS AND LOCATIONS:
Overall Officials: Salih, Prof. Dr., Principal Investigator — CCU Translational Immunology
Locations (1):
- University Hospital Tuebingen, Tübingen, Baden-Würtemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hackenbruch C, Bauer J, Heitmann JS, Maringer Y, Nelde A, Denk M, Zieschang L, Kammer C, Federmann B, Jung S, Martus P, Malek NP, Nikolaou K, Salih HR, Bitzer M, Walz JS. FusionVAC22_01: a phase I clinical trial evaluating a DNAJB1-PRKACA fusion transcript-based peptide vaccine combined with immune checkpoint inhibition for fibrolamellar hepatocellular carcinoma and other tumor entities carrying the oncogenic driver fusion. Front Oncol. 2024 Mar 28;14:1367450. doi: 10.3389/fonc.2024.1367450. eCollection 2024. PMID 38606105